CLINICAL TRIAL: NCT01990833
Title: Molecular Characteristics of the Persistent Intestinal Fistulae After Glue Application
Status: Completed | Type: Observational
Sponsor: Jianan Ren (Other)
Responsible Party: Sponsor-Investigator, Jianan Ren, Vice president, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Other Study IDs: 20120101
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Enterocutaneous Fistulas
MeSH Terms: conditions — Intestinal Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasmas and fistula tissues
Oversight: Data Monitoring Committee: No

SUMMARY:
For non-healing ulcers, abnormal periods of wound healing processes: inflammation, proliferation and remodelling, are believed to lead to chronic wounds. As a chronic "stalled" wound, investigators hypothesized that these glue-assisted closure (GAC)-failed enterocutaneous fistula (ECF) might have a prolonged inflammatory phase modulated by excessive pro-inflammatory cytokines or proteases. The aim of this study was to analyze the chemicals in ECF wounds in order to determine patients' condition and fitness for GAC.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old;
* single tubular (tract length >2 cm) ECF;
* low output volume (<200 ml/24h);

Exclusion Criteria:

* fistulas of cancer-infiltrated;
* associated abscess;
* foreign bodies;
* distal bowel obstruction;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low-output enterocutaneous fistulas receiving glue application
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Fistula closure after glue application | 7 days
  No fistula output